CLINICAL TRIAL: NCT04830085
Title: Factors Associated With Adenomyosis and a Clinical Scoring System for the Diagnosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Hakan Aytan, Professor Dr., Mersin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017/22
Record Dates: First submitted 2021-03-27; First posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-04

CONDITIONS: Adenomyosis
MeSH Terms: conditions — Adenomyosis | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with adenomyosis (Experimental): Hysterectomy (abdominal or vaginal or laparoscopic) Histopathological assessment Adenomyosis was diagnosed with histopathological assessment.
  Interventions: Procedure: Hysterectomy
- Patients without adenomyosis (Active Comparator): Hysterectomy (abdominal or vaginal or laparoscopic) Histopathological assessment Adenomyosis was excluded with histopathological assessment.
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy — Hysterectomy (abdominal, vaginal or laparoscopic)
  Other Names: Histopathological evaluation

SUMMARY:
Adenomyosis is a relatively common benign disorder in which endometrial gland and stroma are located within the myometrium resulting angiogenesis of the spiral vessel, hypertrophy of the surrounding smooth muscles and enlargement of the uterus. So far the definitive diagnosis still requires histologic analysis of the hysterectomy specimens or hysteroscopic or laparoscopic biopsy. There is no specific laboratory tests and reliable clinical standards for the diagnosis. The preoperative diagnosis of adenomyosis, would prevent unnecessary therapies, loss of time and use of resources in vain. Therefore precise prediction of this disease without surgery gains importance. Developing a scoring system with clinical evaluation for this purpose will be very helpful in solving this problem. From this point, the investigators aimed to develop a scoring system that will predict presence of adenomyosis wİth high sensitivity using clinical evaluation methods such as history, physical examination, ultrasonography and laboratory tests. A prospective cohort study was conducted with 221 patients. In the study, the investigators have created a clinical scoring system for this purpose for the first time in the literature. In this scoring system, there are simple parameters that can be easily used by the clinician, have a low cost and are repeatable. The effect of each parameter on predicting adenomyosis is different, and the total effect can be calculated according to the answer to be given to all questions. In this simple scoring system, parity, menarche, VAS scores of dysmenorrhea and dyspareunia, myometrial heterogeneity in ultrasonography and presence of tenderness during pelvic examination were found to be useful parameters in predicting the diagnosis of adenomyosis.

DETAILED DESCRIPTION:
A prospective cohort study was conducted in Mersin University Faculty of Medicine Department of Obstetrics and Gynecology between 10.02.2017 and 10.08.2017 with 221 patients who had undergone hysterectomy for benign disorders. The patients who were admitted to the hospital with the hysterectomy indications for benign pathologies were visited before the operation and a detailed anamnesis was obtained. Physical and pelvic examinations with transvaginal ultrasound examinations were performed by the same investigator. Demographic characteristics, obstetric and gynecologic histories were noted. The amount of percieved pain was measured with Visual Analog Scale (VAS). Observing myometrial cysts, enlarged uterus, heterogeneous myometrium and or focal nodular areas during transvaginal sonography was considered to suggest adenomyosis. The hysterectomy specimes were evaluated by department of pathology. The diagnosis of adenomyosis was based on the presence of glandular extension ≥2.5 mm below the endometrial myometrial interface.

In order to develop a scoring system a regression analysis was carried out to find the parameters that were associated with the presence of adenomyosis. Number of parities, dyspareunia and dysmenorrhea VAS scores, age of menarche, presence of uterine tenderness and detection of heterogenous myometrium and myometrial cysts during ultrasonography were found to be the significant parameters.

ELIGIBILITY:
Inclusion Criteria:

* The patients who were admitted to the hospital with the hysterectomy indications for benign pathologies

Exclusion Criteria:

* Patients with postoperative diagnosis of gynecologic malignancies and who were pregnants

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
Severity of dysmenorrhea measured with Visual Analog Scale | 6 months
Severity of dyspareunia measured with Visual Analog Scale | 6 months
Detection of myometrial heterogeneity during transvaginal ultrasonographic examination | 6 months
Detection of myometrial cysts during transvaginal ultrasonographic examination | 6 months
Presence of uterine tenderness during pelvic examination | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: HAKAN AYTAN, Prof. MD, Study Director — Mersin University
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No